CLINICAL TRIAL: NCT03385252
Title: The Mazira Project: An Evaluation of Eggs During Complementary Feeding in Rural Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Kamuzu University of Health Sciences (Other); Washington University School of Medicine (Other); University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1125193
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Infant Malnutrition
Keywords: complementary feeding; eggs; infant growth; stunting; cognitive development; choline; vitamin B12; microbiome
MeSH Terms: conditions — Infant Nutrition Disorders; Growth Disorders | interventions — Eggs

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will not be masked. Data collectors will not be informed of the participant's group assignments. Data analysis will be conducted on blinded datasets until the primary analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg Group (Experimental): Egg Intervention: Provision of eggs to caregivers of enrolled infants, with instructions to prepare and feed one egg to the infant each day for 6 months time. Households will be visited twice weekly to provide eggs and monitor intake.
  Interventions: Other: Eggs; Behavioral: Visits
- Control Group (Active Comparator): Control Group: Caregivers will receive a food basket at the end of the study. Throughout the trial, households will be visited twice weekly and asked about food intake.
  Interventions: Behavioral: Visits

INTERVENTIONS:
Other: Eggs — Eggs provided as complementary food for the infant
  Arms: Egg Group
Behavioral: Visits — Twice weekly household visits by study staff

SUMMARY:
The Mazira Project is a study of the effect of egg consumption on growth, development and gut health of infants in Malawi. The study randomly assigns infants to receive one egg per day over six months or to receive an equivalent value of food at the end of six months. Growth, achievement of developmental milestones, gut microbiome composition and other measures of nutritional status are compared between the two groups to determine whether regular egg consumption benefits Malawian infants.

DETAILED DESCRIPTION:
The aim of the Mazira Project is to determine whether daily consumption of an egg improves the growth and development of infants in rural Malawi. In Malawi, 37% of children under five years old are stunted, or shorter than expected for their age (1). Most stunting occurs when children are less than 2 years old. Stunting is a sign of long-term undernutrition and is associated with delayed cognitive development. Eggs provide protein, fatty acids, vitamin B12, choline and other nutrients that may support healthy growth and cognitive development. In a previous trial in Ecuador, infants who were provided eggs for daily consumption showed improved growth and lower rates of stunting than infants who were not provided eggs (2).

Investigators are assessing whether children who consume eggs regularly over six months starting when they are 6 to 9 months old have higher height-for-age scores and lower rates of stunting than children who do not consume eggs regularly. Investigators are also assessing whether egg consumption improves Malawian infants' cognitive development. Because gut health is important for good nutrition, they are testing whether eggs have positive effects on measures of gut health and the gut microbiome. Finally, they are exploring the various metabolic pathways by which the nutrients available in eggs may influence infant growth and development.

Participants are individually, randomly assigned to the egg intervention group or the control group. The mothers of infants who are randomly assigned to the egg intervention group receive 14 eggs each week and are asked to feed the infant one egg each day. Extra eggs are provided because sharing of food is common in Malawian households. The mothers of infants who are randomly assigned to the control group receive a package of foods at the end of the study that is equal in value to the eggs. Each mother/infant pair participates in the study for six months.

When infants are enrolled, a baseline assessment is completed. This assessment includes a blood draw plus testing for anemia and malaria, anthropometric measurements, developmental assessments, 24-hour dietary recall interview, infant health history questionnaire. Mothers' heights and weights are also measured, and each mother is asked about socio-economic and demographic indicators and food security in her household. The anthropometric, dietary and development assessments are repeated after 3 months. At the end of the six month study period, anthropometric, dietary and development assessments are repeated, along with another blood draw.

Additional data collected during the course of the study include: repeat 24-hour dietary recalls and monthly stool sample collection among a subsample of 200 children; twice-weekly observations of the index infant's egg consumption in the egg group or short questionnaire about the index infant's most recent meal in the control group; weekly morbidity history and animal source food consumption questionnaire among all infants; and focus groups and key informant interviews about production, availability and consumption of eggs among communities in the study area.

ELIGIBILITY:
Inclusion Criteria:

* Living in catchment area of Lungwena health center, Mangochi District, Malawi during the study enrollment period
* Singleton birth

Exclusion Criteria:

* Egg allergy
* History of anaphylaxis or any serious allergic reaction requiring emergency medical care
* Congenital or chronic condition impacting growth and development or ability to eat eggs
* Severe anemia (hemoglobin < 5 g/dL)
* Mid-upper arm circumference < 12.5 cm or presence of bipedal edema
* Acute illness or injury warranting hospital referral

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 662 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Length-for-age z-score | 6 months after the start of the intervention
  Child's recumbent length, standardized using the World Health Organization growth standards
Stunting | 6 months after the start of the intervention
  Prevalence of length-for-age z-score <-2

SECONDARY OUTCOMES:
Weight-for-age z-score and prevalence of underweight (WAZ<-2) | 6 months after the start of the intervention
Weight-for-length z-score and prevalence of wasting (WLZ<-2) | 6 months after the start of the intervention
Plasma choline concentration | 6 months after the start of the intervention
  Venous blood collection
Plasma amino acid concentrations | 6 months after the start of the intervention
  Venous blood collection
Cognitive development | 6 months after the start of the intervention
  Measured using the Malawi Development Assessment Tool (MDAT), Infant eye-tracking measures of declarative memory, and delayed imitation tasks

OTHER OUTCOMES:
Plasma concentrations of micronutrient biomarkers (iron, zinc, vitamin A, B12) and lipids | 6 months after the start of the intervention
  Venous blood collection
Microbiome: microbial diversity and abundance | Each month for 6 months
  Stool sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Christine P Stewart, PhD, Principal Investigator — University of California, Davis; Lora Iannotti, PhD, Principal Investigator — Washington University School of Medicine; Chessa Lutter, PhD, Principal Investigator — University of Maryland, College Park; Kenneth M Maleta, PhD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- University of Malawi College of Medicine, Mangochi Campus, Mangochi, Malawi

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be posted in a publicly accessible repository on the Open Science Framework website. Publicly shared data will include all the individual participant data that underlie the results in each publication.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The study protocol and statistical analysis plan for the primary outcome analysis will be posted before data analysis begins. Data and analytic code will be posted within 6 months after publication of the primary outcome results.
Access Criteria: Published data will be made publicly accessible. Unpublished data may be requested by contacting the study Principal Investigator.
URL: https://osf.io/vfrg7/

REFERENCES:
- [Background] National Statistical Office (NSO) [Malawi], ICF, Malawi Demographic and Health Survey 2015-16. Zomba, Malawi and Rockville, Maryland, USA: NSO and ICF; 2017.
- [Background] Iannotti LL, Lutter CK, Stewart CP, Gallegos Riofrio CA, Malo C, Reinhart G, Palacios A, Karp C, Chapnick M, Cox K, Waters WF. Eggs in Early Complementary Feeding and Child Growth: A Randomized Controlled Trial. Pediatrics. 2017 Jul;140(1):e20163459. doi: 10.1542/peds.2016-3459. Epub 2017 Jun 7. PMID 28588101
- [Result] Stewart CP, Caswell B, Iannotti L, Lutter C, Arnold CD, Chipatala R, Prado EL, Maleta K. The effect of eggs on early child growth in rural Malawi: the Mazira Project randomized controlled trial. Am J Clin Nutr. 2019 Oct 1;110(4):1026-1033. doi: 10.1093/ajcn/nqz163. PMID 31386106
- [Derived] Werner ER, Haskell MJ, Arnold CD, Caswell BL, Iannotti LL, Lutter CK, Maleta KM, Stewart CP. The Effects of One Egg Per Day on Vitamin A Status Among Young Malawian Children: A Secondary Analysis of a Randomized Controlled Trial. Curr Dev Nutr. 2023 Feb 23;7(3):100053. doi: 10.1016/j.cdnut.2023.100053. eCollection 2023 Mar. PMID 37181936
- [Derived] Werner ER, Arnold CD, Caswell BL, Iannotti LL, Lutter CK, Maleta KM, Stewart CP. The Effects of 1 Egg per Day on Iron and Anemia Status among Young Malawian Children: A Secondary Analysis of a Randomized Controlled Trial. Curr Dev Nutr. 2022 May 13;6(6):nzac094. doi: 10.1093/cdn/nzac094. eCollection 2022 Jun. PMID 35755939
- [Derived] Bragg MG, Prado EL, Arnold CD, Zyba SJ, Maleta KM, Caswell BL, Bennett BJ, Iannotti LL, Lutter CK, Stewart CP. Plasma Choline Concentration Was Not Increased After a 6-Month Egg Intervention in 6-9-Month-Old Malawian Children: Results from a Randomized Controlled Trial. Curr Dev Nutr. 2022 Feb 23;6(2):nzab150. doi: 10.1093/cdn/nzab150. eCollection 2022 Feb. PMID 35233478
- [Derived] Caswell BL, Arnold CD, Lutter CK, Iannotti LL, Chipatala R, Werner ER, Maleta KM, Stewart CP. Impacts of an egg intervention on nutrient adequacy among young Malawian children. Matern Child Nutr. 2021 Jul;17(3):e13196. doi: 10.1111/mcn.13196. Epub 2021 May 11. PMID 33974324
- [Derived] Lutter CK, Caswell BL, Arnold CD, Iannotti LL, Maleta K, Chipatala R, Prado EL, Stewart CP. Impacts of an egg complementary feeding trial on energy intake and dietary diversity in Malawi. Matern Child Nutr. 2021 Jan;17(1):e13055. doi: 10.1111/mcn.13055. Epub 2020 Jul 20. PMID 33128502
- [Derived] Prado EL, Maleta K, Caswell BL, George M, Oakes LM, DeBolt MC, Bragg MG, Arnold CD, Iannotti LL, Lutter CK, Stewart CP. Early Child Development Outcomes of a Randomized Trial Providing 1 Egg Per Day to Children Age 6 to 15 Months in Malawi. J Nutr. 2020 Jul 1;150(7):1933-1942. doi: 10.1093/jn/nxaa088. PMID 32286620